CLINICAL TRIAL: NCT06270693
Title: Effect of Endodontic Treatment on Serum High Sensitivity C-reactive Protein and Complete Hemogram Indices in Patients With Cardiovascular Disease With and Without Apical Periodontitis: A Prospective Interventional Study
Brief Title: hsCRP & CH Indices in Patients With Coronary Artery Disease With and Without Apical Periodontitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dr Sushma
Record Dates: First submitted 2024-01-13; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Apical Periodontitis; Coronary Artery Disease
Keywords: apical periodontitis; coronary artery disease
MeSH Terms: conditions — Periapical Periodontitis; Coronary Artery Disease | interventions — Endodontics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAD WITH AP (Experimental): CORONARY ARTERY DISEASE WITH APICAL PERIODONTITIS
  Interventions: Procedure: Endodontic treatment
- CAD WITHOUT AP (No Intervention): CORONARY ARTERY DISEASE WITHOUT AP

INTERVENTIONS:
Procedure: Endodontic treatment — Root canal treatment
  Arms: CAD WITH AP

SUMMARY:
Endodontic treatment is done in Patients with chronic pulp exposure in patients with Coronary Artery Disease and systemic inflammatory markers recorded before and and after treatment and compared with patients with Coronary Artery Disease without chronic pulp exposure.

DETAILED DESCRIPTION:
Endodontic treatment is done in Patients with chronic pulp exposure in patients with Coronary Artery Disease and systemic inflammatory markers recorded before and and after treatment and compared with patients with Coronary Artery Disease without chronic pulp exposure. Systemic inflammatory burden is assessed before and after endodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Coronary artery disease patients with and without chronic pulp exposure

Exclusion Criteria:

* Other systemic diseases
* Antibiotics for More than 1 month
* Smoking
* Analgesics more than 1 week

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Serum hsCRP | 12 months
  Systemic inflammatory burden assessed
complete hemogram indices | 12 months
  Systemic inflammatory burden assessed

SECONDARY OUTCOMES:
Periapical index SCORE CHANGE | 12 months
  1-5 ordinal scale,5 worse outconpme & HEALING ASSESSED

CONTACTS AND LOCATIONS:
Overall Officials: DR SANJAY TEWARI, MDS, Study Director — Post Graduate Institute Of Dental Sciences,Rohtak
Locations (1):
- PGIDS, Rohtak, Haryana, India